CLINICAL TRIAL: NCT06416748
Title: Minimally Invasive Simple Hysterectomy in Low Risk Cervical Cancer
Acronym: LASH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Bizzarri Nicolò, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAcc & SHape - LASH trial
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cervical Cancer; Cervix Cancer
Keywords: Cervical cancer; Minimally invasive surgery in cervical cancer; Robotic surgery in cervical cancer; Laparoscopic surgery in cervical cancer; LACC trial; SHAPE trial; Low risk cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with SHAPE inclusion criteria (FIGO 2018 stage IA2 and IB1 up to 2 cm, with limited stromal invasion: < 10 mm on LEEP/cone and < 50% depth on imaging) should undergo conization with surgical margins free from invasive disease or conization with involved surgical margins followed by MRI scan or expert ultrasound scan showing no residual disease. In case of residual disease at post conization imaging still fitting inclusion criteria, another conization is recommended. After these steps minimally invasive (laparoscopy or robotic) simple hysterectomy is performed with sentinel lymph node biopsy algorithm. Adjuvant therapy is given only in case of positive surgical margins, metastatic lymph nodes, and extensive LVSI with depth of stromal infiltration >2/3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): Patients with SHAPE inclusion criteria (FIGO 2018 stage IA2 and IB1 up to 2 cm, with limited stromal invasion: < 10 mm on LEEP/cone and < 50% depth on imaging) should undergo conization with surgical margins free from invasive disease or conization with involved surgical margins followed by MRI scan or expert ultrasound scan showing no residual disease. In case of residual disease at post conization imaging still fitting inclusion criteria, another conization is recommended. After these steps minimally invasive (laparoscopy or robotic) simple hysterectomy is performed with sentinel lymph node biopsy algorithm. Adjuvant therapy is given only in case of positive surgical margins, metastatic lymph nodes, and extensive LVSI with depth of stromal infiltration over 2/3.
  Interventions: Procedure: Minimally invasive simple hysterectomy

INTERVENTIONS:
Procedure: Minimally invasive simple hysterectomy — Patients with SHAPE inclusion criteria (FIGO 2018 stage IA2 and IB1 up to 2 cm, with limited stromal invasion: < 10 mm on LEEP/cone and < 50% depth on imaging) should undergo conization with surgical margins free from invasive disease or conization with involved surgical margins followed by MRI scan or expert ultrasound scan showing no residual disease. In case of residual disease at post conization imaging still fitting inclusion criteria, another conization is recommended. After these steps minimally invasive (laparoscopy or robotic) simple hysterectomy is performed with sentinel lymph node biopsy algorithm. Adjuvant therapy is given only in case of positive surgical margins, metastatic lymph nodes, and extensive LVSI with depth of stromal infiltration over 2/3.
  Other Names: simple hysterectomy

SUMMARY:
The rationale of the present study is to assess the safety of the minimally invasive surgery approach in patients meeting the SHAPE trial inclusion criteria.The SHAPE trial was designed to answer the clinical question of whether simple hysterectomy could be performed instead of radical hysterectomy in low-risk early stage cervical cancer but not the surgical approach. The favorable oncological outcome observed in SHAPE despite 75% of patients were treated with minimally invasive approach suggests that this approach may be safe. However, the trial was not designed to analyze oncological outcomes from surgical approach.

DETAILED DESCRIPTION:
The Laparoscopic Approach to Cervical Cancer (LACC) Trial showed that minimally invasive radical hysterectomy was associated with lower rates of disease-free survival and overall survival than open abdominal radical hysterectomy among women with early-stage cervical cancer. Since then, the standard of care in terms of surgical approach to radical hysterectomy has been considered the laparotomy. More recently, the SHAPE trial results were presented showing that in patients with low-risk cervical cancer (defined as FIGO 2018 stage IA2 and IB1 up to 2 cm, with limited stromal invasion: < 10 mm on LEEP/cone and < 50% depth on MRI) simple hysterectomy was not inferior to radical hysterectomy for what concerned pelvic recurrence, with less complications and better quality of life. However, SHAPE trial was not designed to assess the surgical approach.

The rationale of the present study is to assess the safety of the minimally invasive surgery approach in patients meeting the SHAPE trial inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma of uterine cervix
* FIGO 2018 stage IA2-IB1 (≤2cm) with depth of infiltration ≤10mm on conization specimen
* FIGO 2018 stage IA2-IB1 (≤2cm) with depth of infiltration ≤50% at pre-conization MRI-scan or "expert" US-scan.
* Age ≥18 years

Exclusion Criteria:

* Neuroendocrine, clear cell, serous carcinoma
* Depth of infiltration >10 mm on conization specimen
* Depth of infiltration >50% at pre-conization imaging
* Cervical tumor >2 cm
* Diagnosis on inadvertent hysterectomy
* Neoadjuvant chemotherapy
* Previous pelvic radiotherapy
* Pregnant women
* Contraindications to surgery
* Lymph nodes >15 mm short axis
* Fertility sparing treatment or desire
* Recurrent cervical cancer
* Time between cervical cancer diagnosis and hysterectomy >4 months if conization with tumor negative margins
* Time between cervical cancer diagnosis and hysterectomy >3 months if conization with invasive tumor positive margins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients meeting the inclusion criteria
Enrollment: 974 (Estimated)
Dates: Start 2024-10-27 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
3-year DFS | 36 months after surgery
  disease free survival at 3 years

SECONDARY OUTCOMES:
3-year recurrence rate (including pelvic recurrence rate) | 36 months after surgery
3-year overall survival | 36 months after surgery
intra-operative and post-operative complications | 36 months after surgery
Rate of upstage after surgery | 36 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nicolò Bizzarri, MD, Study Director — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Giovanni Scambia, Prof., Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Denis Querleu, Prof., Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Francesco Fanfani, Prof., Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Anna Fagotti, Prof., Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Gabriella Ferrandina, Prof., Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Valerio Gallotta, MD, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Luigi Pedone Anchora, MD, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Result] Plante M, Kwon JS, Ferguson S, Samouelian V, Ferron G, Maulard A, de Kroon C, Van Driel W, Tidy J, Williamson K, Mahner S, Kommoss S, Goffin F, Tamussino K, Eyjolfsdottir B, Kim JW, Gleeson N, Brotto L, Tu D, Shepherd LE; CX.5 SHAPE investigators; CX.5 SHAPE Investigators. Simple versus Radical Hysterectomy in Women with Low-Risk Cervical Cancer. N Engl J Med. 2024 Feb 29;390(9):819-829. doi: 10.1056/NEJMoa2308900. PMID 38416430
- [Result] Ramirez PT, Frumovitz M, Pareja R, Lopez A, Vieira M, Ribeiro R, Buda A, Yan X, Shuzhong Y, Chetty N, Isla D, Tamura M, Zhu T, Robledo KP, Gebski V, Asher R, Behan V, Nicklin JL, Coleman RL, Obermair A. Minimally Invasive versus Abdominal Radical Hysterectomy for Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1895-1904. doi: 10.1056/NEJMoa1806395. Epub 2018 Oct 31. PMID 30380365
- [Derived] Bizzarri N, Querleu D, Ramirez PT, Plante M, Giannarelli D, Falconer H, Abu-Rustum NR, Cibula D, Martinez A, Laas E, Fotopoulou C, Chiva L, Pavone M, Pedone Anchora L, Fanfani F, Fagotti A, Scambia G. Minimally invasive simple hysterectomy in low-risk cervical cancer: a single-arm trial with stopping rules (ENGOT-cx23/MITO/LASH trial). Int J Gynecol Cancer. 2025 Jun;35(6):101818. doi: 10.1016/j.ijgc.2025.101818. Epub 2025 Apr 5. PMID 40328196